CLINICAL TRIAL: NCT03113539
Title: Low-dose, EKG-gated CT Validity for the Evaluation of Ascendant Aortic Aneurysm.
Brief Title: Low-dose Gated CT Validity for the Evaluation of Ascendant Aortic Aneurysm.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Paul Farand, MD, FRCPC, Professeur agréé, Directeur du service de cardiologie, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-1074
Record Dates: First submitted 2017-04-02; First posted 2017-04-13 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Ascendant Aortic Aneurysm
MeSH Terms: interventions — Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects awaiting for an aortic evaluation (Experimental): Subjects already waiting for an aortic evaluation, either a first diagnostic scan or follow-up of a known aneurysm.
  Each subjects will have the two CT-scans on the same day.
  Interventions: Other: Modified Low-dose, EKG-gated CT without contrast for the evaluation of aortic aneurysm

INTERVENTIONS:
Other: Modified Low-dose, EKG-gated CT without contrast for the evaluation of aortic aneurysm — On the same day, the subject will do :
  1. Modified low-dose, EKG-gated CT without contrast
  2. Usual high-dose, EKG-gated CT with contrast
  Comparing aortic diameters from the two protocols.

SUMMARY:
We will demonstrate the validity of measurements with a low-dose, EKG-gated CT without contrast in the ascending aorta evaluation, compared with the current Angio-CT measurements.

DETAILED DESCRIPTION:
The actual protocol used in aorta evaluation consist of two CT-scans on the same study. The first scan that detects calcifications is using parameters with low-dose current, non EKG-gated and without contrast. The second scan uses iodine-contrast, EKG-gating and higher current dose to obtain higher image quality of diagnostic value.

The study will optimize the first scan parameters and compare the measures of the aorta diameters from the standard protocol.

By modifying the first scan parameters, we would demonstrate that the follow-up of an aortic aneurysm can safely be made with lower radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old and more
* 85 bpm or less

Exclusion Criteria:

* aortic material
* EKG gating not possible
* aorta pathology (thrombus, dissection)

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Measures validity (aorta diameter in mm from scan images) | 12 months
  Comparing aorta diameters from the two modalities.

SECONDARY OUTCOMES:
Radiation (in msev from scanner report) | 12 months
  Comparing radiation exposure with the two modalities

CONTACTS AND LOCATIONS:
Overall Officials: Paul Farand, Principal Investigator — Université de Sherbrooke
Locations (1):
- Sherbrooke University Hospital, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No